CLINICAL TRIAL: NCT00966953
Title: Development of Clinical Method to Determination Triclosan Retention in Plaque Following Brushing.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: William DeVizio/VP - Clinical Research, Colgate Palmolive
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ERO-0907-PLA-16-RR
Record Dates: First submitted 2008-09-26; First posted 2009-08-27 (Estimated); Results first posted 2009-08-27 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Gingival Diseases
MeSH Terms: conditions — Gingival Diseases | interventions — Fluorides; Triclosan; honokiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fluoride Toothpaste (Placebo Comparator): fluoride control
  Interventions: Drug: Fluoride
- Total/Whitening (Active Comparator): positive control
  Interventions: Drug: Triclosan/Fluoride toothpaste
- antibacterial plant extract 1 (Experimental): Honokiol
  Interventions: Drug: Fluoride
- antibacterial plant extract 2 (Experimental): magnolol
  Interventions: Drug: Fluoride; Other: antibacterial plant extract

INTERVENTIONS:
Drug: Fluoride — Brush twice daily
  Arms: Fluoride Toothpaste
Drug: Triclosan/Fluoride toothpaste — Brush twice daily
  Arms: Total/Whitening
Drug: Fluoride — Brush twice daily
  Other Names: honokiol
  Arms: antibacterial plant extract 1
Drug: Fluoride — Brush twice daily
  Arms: antibacterial plant extract 2
Other: antibacterial plant extract — Brush twice daily
  Other Names: Honokiol
  Arms: antibacterial plant extract 2

SUMMARY:
Clinical research study to determine the anti-plaque efficacy of prototype dentifrices via a 4-day brushing regiment

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers 18-65 years of age.
* Good general health.
* Must sign informed consent form.
* Must discontinue oral hygiene on the mornings of each appointment and between sampling periods.
* No history of allergy to personal care consumer products, or their ingredients, relevant to any ingredient in the test products as determined by the dental/medical professional monitoring the study.

Exclusion Criteria:

* Medical condition which requires pre-medication prior to dental procedures/visits.
* Medical condition which precludes eating/drinking for 12 hrs.
* History of allergy to common dentifrice ingredients.
* Subjects unable or unwilling to sign the informed consent form.
* Moderate or advanced periodontal disease.
* Two or more decayed untreated dental sites at screening.
* Other disease of the hard or soft oral tissues.
* Impaired salivary function (e.g. Sjogren's syndrome or head and neck irradiation).
* Use of medications that can currently affect salivary flow.
* Current use of antibiotics.
* Use of antibiotics or antimicrobial drugs within 30 days prior to study visit #1.
* Pregnant or nursing women.
* Participation in any other clinical study within 30 days prior to enrollment into this study.
* Use of tobacco products.
* Subjects who must receive dental treatment during the study dates.
* Current use of Antibiotics for any purpose.
* Immune compromised individuals (HIV,AIDS, immuno suppressive drug therapy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanfang Ren, DDS, Principal Investigator
Locations (1):
- Eastman Dental Center - University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The dental clinic staff recruited for this study.
Groups:
- Fluoride Control, Magnolol,Total/Whitening,Honokiol: 1st-fluoride only control,2nd-fluoride/magnolol,3rd-triclosan/fluoride control, 4th-fluoride/honokiol
- Total/Whitening, Honokiol, Fluoride Control, Magnolol: 1st-triclosan/fluoride control, 2nd-fluoride/honokiol, 3rd-fluoride only control,4th-fluoride/magnolol
- Honokiol, Fluoride Control, Magnolol, Total/Whitening: 1st-fluoride/honokiol, 2nd-fluoride only control, 3rd-fluoride/magnolol,4th-triclosan/fluoride control
- Magnolol, Total/Whitening, Honokiol, Fluoride Control: 1st-fluoride/Magnolol, 2nd-Fluoride/triclosan control, 3rd-fluoride/Honokiol,4th-fluoride only control
Period: 1st Intervention
Arm/Group | Fluoride Control, Magnolol,Total/Whitening,Honokiol | Total/Whitening, Honokiol, Fluoride Control, Magnolol | Honokiol, Fluoride Control, Magnolol, Total/Whitening | Magnolol, Total/Whitening, Honokiol, Fluoride Control
Started | 6 | 6 | 6 | 7
Completed | 6 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: 1 Week Washout After 1st Intervention
Arm/Group | Fluoride Control, Magnolol,Total/Whitening,Honokiol | Total/Whitening, Honokiol, Fluoride Control, Magnolol | Honokiol, Fluoride Control, Magnolol, Total/Whitening | Magnolol, Total/Whitening, Honokiol, Fluoride Control
Started | 6 | 6 | 6 | 7
Completed | 6 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: 2nd Intervention
Arm/Group | Fluoride Control, Magnolol,Total/Whitening,Honokiol | Total/Whitening, Honokiol, Fluoride Control, Magnolol | Honokiol, Fluoride Control, Magnolol, Total/Whitening | Magnolol, Total/Whitening, Honokiol, Fluoride Control
Started | 6 | 6 | 6 | 7
Completed | 6 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: 1 Week Washout After 2nd Intervention
Arm/Group | Fluoride Control, Magnolol,Total/Whitening,Honokiol | Total/Whitening, Honokiol, Fluoride Control, Magnolol | Honokiol, Fluoride Control, Magnolol, Total/Whitening | Magnolol, Total/Whitening, Honokiol, Fluoride Control
Started | 6 | 6 | 6 | 7
Completed | 6 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: 3rd Intervention Order
Arm/Group | Fluoride Control, Magnolol,Total/Whitening,Honokiol | Total/Whitening, Honokiol, Fluoride Control, Magnolol | Honokiol, Fluoride Control, Magnolol, Total/Whitening | Magnolol, Total/Whitening, Honokiol, Fluoride Control
Started | 6 | 6 | 6 | 7
Completed | 6 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: 1 Week Washout After 3rd Intervention
Arm/Group | Fluoride Control, Magnolol,Total/Whitening,Honokiol | Total/Whitening, Honokiol, Fluoride Control, Magnolol | Honokiol, Fluoride Control, Magnolol, Total/Whitening | Magnolol, Total/Whitening, Honokiol, Fluoride Control
Started | 6 | 6 | 6 | 7
Completed | 6 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: 4th Intervention Order
Arm/Group | Fluoride Control, Magnolol,Total/Whitening,Honokiol | Total/Whitening, Honokiol, Fluoride Control, Magnolol | Honokiol, Fluoride Control, Magnolol, Total/Whitening | Magnolol, Total/Whitening, Honokiol, Fluoride Control
Started | 6 | 6 | 6 | 7
Completed | 6 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoride Control, Magnolol,Total/Whitening,Honokiol | Total/Whitening, Honokiol, Fluoride Control, Magnolol | Honokiol, Fluoride Control, Magnolol, Total/Whitening | Magnolol, Total/Whitening, Honokiol, Fluoride Control | Total
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 7 | 25
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42 (11.8) | 37.8 (11.6) | 46.4 (10.9) | 44.3 (7) | 42.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 7 | 15
  Male | 4 | 3 | 3 | 0 | 10
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Plaque Index
Description: Plaque score scale: Units on a scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque, 3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Fluoride Only: Control toothopaste
- Total/Whitening: Control toothpaste
- Herbal Extract Toothpaste: Fluoride/Honokiol extract toothpaste
- Herbal Extract Toothpaste: Fluoride/Magnolol extract toothpaste
Arm/Group | Fluoride Only | Total/Whitening | Herbal Extract Toothpaste | Herbal Extract Toothpaste
Number analyzed (Participants) | 25 | 25 | 25 | 25
Units on a scale | 2.45 (0.47) | 2.22 (0.46) | 2.54 (0.44) | 2.56 (0.46)
Statistical Analysis 1: Comparison: Fluoride Only vs Total/Whitening vs Herbal Extract Toothpaste vs Herbal Extract Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANOVA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days